CLINICAL TRIAL: NCT01109875
Title: Screening for Fabry Disease Among Young Stroke Patients in an Israeli Stroke Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Yair Lampl, Professor Yair Lampl, Wolfson Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Fabry Disease in the Young Stroke
MeSH Terms: interventions — Hematologic Tests

INTERVENTIONS:
Other: blood test — Dry blood spots (DBS) analysis of a- galactosidase-A activity will be used for male patients' diagnosis. Males and females with enzymatic activity bellow the test's cut-off will be further diagnosed by gene sequencing. Since females are heterozygote and may have high residual levels of active enzyme, female patients with a- galactosidase-A activity of 30% bellow averaged normal range will also be further diagnosed by gene sequencing as described before (8).

SUMMARY:
The purpose of this study is to determine the incidence of Fabry Disease in young stroke patients in an Israeli stroke clinic.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of stoke or TIA Time period within last 5 years -

Exclusion Criteria:

Known diagnosis of stroke or index event due to trauma

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-05; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
positive screening of fabry disease | past 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Dept. Edith Wolfson Medical Center, Holon, Israel